CLINICAL TRIAL: NCT01067170
Title: The Effect of Pneumatic Compression Stockings on Hemodynamic Parameters in Hemodialysis Patients: A Randomized Crossover Trial
Brief Title: Pneumatic Compression Stockings During Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Dr Jennifer MacRae, Director, Hemodialysis and Vascular Access, University of Calgary
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: E-21937
Record Dates: First submitted 2010-02-09; First posted 2010-02-11 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2012-12

CONDITIONS: Hemodialysis
Keywords: Hemodialysis; Intradialytic hypotension
MeSH Terms: interventions — Intermittent Pneumatic Compression Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pneumatic compression stockings (Experimental)
  Interventions: Device: Pneumatic Compression Stockings

INTERVENTIONS:
Device: Pneumatic Compression Stockings — Thigh-high pneumatic compression stockings

SUMMARY:
This study aims to determine the effect of pneumatic compression devices (PCDs) on central blood volume in hemodialysis patients. We hypothesize that PCDs will help maintain central blood volume, and therefore prevent sudden decreases in blood pressure during hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* on hemodialysis at least 3 months
* on hemodialysis at least 3 times per week

Exclusion Criteria:

* dialyzing with a central venous catheter
* vascular access dysfunction
* peripheral vascular disease
* active medical issue
* unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2008-11; Primary Completion 2011-02 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Central blood volume | pre and post hemodialysis

SECONDARY OUTCOMES:
cardiac output | pre and post hemodialysis
cardiac index | pre and post hemodialysis
systemic vascular resistance | pre and post hemodialysis
intracellular fluid volume | pre and post hemodialysis
extracellular fluid volume | pre and post hemodialysis
total body water | pre and post hemodialysis

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer M MacRae, MD MSc, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

REFERENCES:
- [Result] Tai DJ, Ahmed SB, Palacios-Derflingher L, Hemmelgarn BR, MacRae JM; Alberta Kidney Disease Network. Pneumatic compression devices during hemodialysis: a randomized crossover trial. Nephrol Dial Transplant. 2013 Apr;28(4):982-90. doi: 10.1093/ndt/gfs502. Epub 2012 Nov 7. PMID 23136215